CLINICAL TRIAL: NCT03463798
Title: Assesment of New Devices for the Diagnostic Evaluation of Diaphragmatic Dysfunction
Acronym: DYSDIA
Status: Completed | Type: Observational
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03665-48
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Diaphragmatic Paralysis; Healthy Volunteers
Keywords: structured light plethysmography; sonar; transdiaphragmatic pressure
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with a suspicion of diaphragmatic dysfunction
  Interventions: Device: Sonar; Device: Structured light plethysmography (SLP)
- Healthy volunteers: Subjects without any medical condition
  Interventions: Device: Sonar; Device: Structured light plethysmography (SLP)

INTERVENTIONS:
Device: Sonar — Measurements of chest wall and abdominal wall movement will be performed while subjects are breathing quietly
Device: Structured light plethysmography (SLP) — Measurements of chest wall and abdominal wall movement will be performed while subjects are breathing quietly

SUMMARY:
this study aim to evaluate wether new, non-invasive and non-contact devices such as Structured Light Plethysmography (SLP) and Sonar would be able to accurately detect and quantify diaphragm dysfunction (mono-or-bilateral) by assessing the asymmetric chest wall motion generated during spontaneous breathing as compared with a classic, standard and invasive technique.

DETAILED DESCRIPTION:
The measurements of chest and abdominal wall movements during quiet tidal breathing will be performed simultaneously using SLP and Sonar devices.

Subjects will be asked to sit down on a chair with their neck in a neutral position and their back as straight as possible. The SLP and the Sonar will be lined up to project the grid of light and the ultrasonic wave sonar over the participant's chest and abdomen. Data will be collected during 5 minutes of tidal breathing. The same procedure will be repeated while having the patient lying down in supine position on the same chair for 5 additional minutes. During both sessions (sitting and supine), patients will be asked to perform a gentle inspiratory capacity (IC) maneuver to better appreciate the thoraco-abdominal asymmetry and distortion.

ELIGIBILITY:
FOR HEALTHY VOLUNTEERS

Inclusion Criteria:

* no respiratory disease
* no neurologic disease
* no thoracic deformation

Exclusion criteria

* respiratory disease
* neurologic disease
* thoracic deformation

FOR PATIENTS

Inclusion Criteria:

* patients with a suspicion of diaphragmatic dysfunction

Exclusion Criteria:

* pregnant women
* contraindications to standard procedure requiring transdiaphragmatic measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a suspicion of diaphragmatic dysfunction and healthy volunteers without any medical condition.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
amplitude of displacement of thoraco-abdominal compartments | 10 minutes
  asymmetry of displacement of thoraco-abdominal compartments during tidal breathing and respiratory manoeuvres

SECONDARY OUTCOMES:
displacement speed of thoraco-abdominal compartments | 10 minutes
  asynchrony of displacement of thoraco-abdominal compartments during tidal breathing and respiratory manoeuvres measurement

CONTACTS AND LOCATIONS:
Overall Officials: Pierantonio LAVENEZIANA, MD, PhD, Principal Investigator — UMRS_1158
Locations (1):
- INSERM-UPC UMR_S 1158 Service de Pneumologie et Réanimation, R3S, Groupe Hospitalier Pitié-Salpêtrière, Paris, France